CLINICAL TRIAL: NCT05429450
Title: Comparative Study on the Efficacy of Periocular Methotrexate Versus Periocular Triamcinolone Injections in Management of Thyroid Associated Orbitopathy
Brief Title: Thyroid Associated Orbitopathy Treatment by Methotrexate Against Triamcinolone Periocular Injections
Acronym: TOMATO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Islam Youssef Swaify, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MD-139-2020
Record Dates: First submitted 2022-06-18; First posted 2022-06-23 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Thyroid Associated Orbitopathy
Keywords: Thyroid associated orbitopathy; Grave's orbitopathy; Periocular injections; Methotrexate; Triamcinolone
MeSH Terms: interventions — Methotrexate; Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Methotrexate (Experimental): Periocular injections of methotrexate
  Interventions: Drug: Methotrexate
- Triamcinolone acetonide (Active Comparator): Periocular injections of triamcinolone acetonide
  Interventions: Drug: Triamcinolone Acetonide

INTERVENTIONS:
Drug: Methotrexate — Three periocular injections of methotrexate at week 0, week 3 and week 6.
  Arms: Methotrexate
Drug: Triamcinolone Acetonide — Three periocular injections of triamcinolone acetonide at week 0, week 3 and week 6.
  Arms: Triamcinolone acetonide

SUMMARY:
The study objective is to investigate the efficacy and safety of periocular injections of methotrexate in management of patients with active moderate to severe thyroid associated orbitopathy in comparison to periocular injections of triamcinolone acetonide.

DETAILED DESCRIPTION:
Recruited subjects will be randomized such that one orbit receives 3 periocular injections of methotrexate and the contralateral orbit receives 3 periocular injections of triamcinolone acetonide at day 0, week 3 and week 6. All study subjects will be followed up for 6 months where outcome measures are assessed at 2 weeks, 1month, 3 months and 6 months after last injection

ELIGIBILITY:
Inclusion Criteria:

1. Bilateral moderate to severe thyroid associated orbitopathy.
2. Clinical Activity score (CAS) ≥ 3.
3. Duration of thyroid associated orbitopathy < 2 years

Exclusion Criteria:

1. Sight threatening thyroid associated orbitopathy (dysthyroid optic neuropathy or exposure keratopathy) in any eye.
2. Glaucoma patients or those known to be steroid responders
3. Presence of orbital infections or any infection in nearby structures as paranasal sinusitis or dental abscess
4. Pregnancy
5. Previous orbital or lid surgeries
6. History of steroid therapy (oral, intravenous or periocular) or other immunosuppressive therapy within the previous 3 months

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
Change in clinical activity score (CAS) | 2 weeks, 1 month, 3 months and 6 months
  Mean change in clinical activity score from baseline. CAS is a 10-point score (0-10) with disease considered active if CAS is >3.

SECONDARY OUTCOMES:
Change in proptosis | 2 weeks, 1 month, 3 months and 6 months
  Mean change in proptosis measured in millimeters by an exopthalmometer compared to baseline proptosis
Change in lid aperture | 2 weeks, 1 month, 3 months and 6 months
  Mean change in lid aperture (distance between upper and lower lid margin measured in millimeters by a ruler
Percentage of overall responders | 3 months and 6 months
  A participant is considered an overall responder if 2 or more of the following:
  1. Improvement of CAS ≥ 2 points.
  2. Improvement of proptosis ≥ 2 mm.
  3. Improvement of lid aperture ≥ 2 mm.
  4. Improvement of soft tissue signs ≥ 1 grade
  5. Improvement of EOM ductions

CONTACTS AND LOCATIONS:
Overall Officials: Haytham E. Nasr, Study Chair — Cairo University; Rania A. El Essawy, Study Director — Cairo University; Kareem B. Elessawy, Study Director — Cairo University; Islam Y. Swaify, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No